CLINICAL TRIAL: NCT05782998
Title: MSCT Measurements of the Lumbar Spinal Canal Regarding Age and Sex.
Brief Title: Normal Range of Measurement of Lumbar Spinal Canal in MSCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yomna Gamal Abozeid, Principal investigator, Assiut University
Other Study IDs: Measurement of spinal canal
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Lumbar Spinal Canal Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study aims to establish a normal range of measurements of lumbar spinal canal.

DETAILED DESCRIPTION:
The knowledge of normal diameter of lumbar spinal canal is very important for diagnosing lumbar spinal canal stenosis and also for performing spinal surgeries at the lumbar level by Neurosurgeons and Orthopedicians. However, it varies widely among ethnic groups and between sexes in the same ethnic group . Spinal canal stenosis (defined as the narrowing of central spinal canal) is a condition in which the anteroposterior (AP) and lateral dimensions of the bony spinal canal are less than normal for corresponding age and sex. Back pain is the commonest manifestation of lumbar canal stenosis which usually results from lumbar spondylosis. Lumber lordosis is a problem of adults, but is now being increasingly seen in youth, probably due to lifestyle changes. Multiple factors play a role in spondylosis, but if it is associated with spinal canal stenosis, its management differs. Radiological evaluation forms an important part in the evaluation and management of lumbar spondylosis. But it requires clear understanding of the normal dimensions of lumbar vertebrae for particular age & sex . Multislice computed tomography (MSCT) scans provides a noninvasive, non-operator dependent method of direct imaging of the spinal canal without injection of intra thecal contrast and is better than MRI for bony detail as in osteophytes. Though there is a wide variation in the capacity of spinal canal in patients who are clinically and radiologically normal. It is said that those with smaller canals are more likely to have symptoms from nerve root compression . By determining normal ranges of spinal canal diameter investigators can make early diagnosis in individuals who have lower diameters of spinal canal. These individuals are predisposed to spinal canal stenosis, which is a major cause of spinal radiculopathies. The recent use of CT for the measurements of the vertebral dimensions such as canal diameter and vertebral dimension has led to better evaluation of vertebral morphometry as compared with x-ray and cadaveric studies . CT scan measurement of lumbar spine demonstrated a mean AP canal diameter between 12 mm and 14 mm with a measurement of 11.5 mm considered small. On CT scan, electronic measurement of the sagittal diameter of the normal bony canal is 11.5 mm . These differences in dimension of the spinal canal across studies demands necessity of study of dimension of the spinal canal in every ethnic group.

ELIGIBILITY:
Inclusion Criteria:

* Normal population without any known vertebral column pathology or complaints in both sex & different age groups.
* Patient fit for CT examination.

Exclusion Criteria:

* Pregnancy.
* Patients having sciatic pain with or without pain in the back.
* Patient having past history of back surgery.
* Patients with osteophytes or developmental anomalies, trauma vertebral fracture and known case of lordosis, scoliosis or kyphosis or other abnormalities in lumbar vertebrae.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Normal population without any known vertebral column pathology or complaints in both sex & different age groups and fit for CT examination.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
MSCT Measurements of the Lumbar Spinal Canal | baseline
  Establish a normal range of measurements of lumbar spinal canal regarding age and sex in Egyptian population.

REFERENCES:
- See also: 1.Spinal Canal measurement at the level of lower three lumbar vertebrae by 128- Slice CT Scanner in Bangladeshi population .Siraj N,Ghafoor N,Parven JP,Deepa KP,Haque MZ.Ibrahim Card Med J 2021 :11 (1):8-13. — https://doi.org/10.3329/icmj.v11i1.58699